CLINICAL TRIAL: NCT01301898
Title: Randomized, Single-blind, Active-controlled, Phase 1/2 Study to Evaluate the Safety and Efficacy of GC1111 (Recombinant Human Iduronate-2-sulfatase) in Hunter Syndrome (Mucopolysaccharidosis II) Patients
Brief Title: To Evaluate the Safety and Efficacy of GC1111 (Recombinant Human Iduronate-2-sulfatase) in Hunter Syndrome Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GC1111_P1/2
Record Dates: First submitted 2011-02-22; First posted 2011-02-23 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Mucopolysaccharidosis II
Keywords: Hunter syndrome; MPS II; Idursulfase
MeSH Terms: conditions — Mucopolysaccharidosis II; Sudden Infant Death

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GC1111_0.5mg/kg (Experimental)
  Interventions: Drug: GC1111_0.5mg/kg
- GC1111_1.0mg/kg (Experimental)
  Interventions: Drug: GC1111_1.0mg/kg
- Elaprase_0.5mg/kg (Active Comparator)
  Interventions: Drug: Elaprase_0.5mg/kg

INTERVENTIONS:
Drug: GC1111_0.5mg/kg
  Arms: GC1111_0.5mg/kg
Drug: GC1111_1.0mg/kg
  Arms: GC1111_1.0mg/kg
Drug: Elaprase_0.5mg/kg
  Arms: Elaprase_0.5mg/kg

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of GC1111 (recombinant human iduronate-w-sulfatase) in Hunter Syndrome (Mucopolysaccharidosis II) patients

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diagnosis of MPS II based on both clinical and biochemical criteria
2. Male, ages 6 to 35 years old
3. Patients who are able to comply with the study requirements
4. Patients who have given voluntary written consent to participate in the study
5. Patients who is acceptable for using an appropriate method of contraception

Exclusion Criteria:

1. History of a tracheostomy or a bone marrow transplant
2. Known hypersensitivity to idursulfase
3. Known shock to idursulfase
4. History of receiving treatment with another investigational therapy within the past 30 days
5. History of a stem cell transplant
6. Known hypersensitivity to any of the components of idursulfase
7. Female

Ages: 6 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2010-05; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Primary Outcome | baseline, every 4 weeks
  measurement of % change of Urine GAG

SECONDARY OUTCOMES:
Secondary Outcome | baseline, every 12 weeks
  * Measurements of the six-minute-walk test (6-MWT)
  * Measurements of liver volume
  * Measurements of heart size and heart function
  * Measurements of joint range of motion
  * Measurements of urine GAG levels
  * Measurements of pulmonary function
  * Evaluate the safety: vital signs, physical examination, laboratory tests, adverse events, immunogenecity

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Irwon-dong, Gangnam-Gu, South Korea

REFERENCES:
- [Derived] Sohn YB, Cho SY, Park SW, Kim SJ, Ko AR, Kwon EK, Han SJ, Jin DK. Phase I/II clinical trial of enzyme replacement therapy with idursulfase beta in patients with mucopolysaccharidosis II (Hunter syndrome). Orphanet J Rare Dis. 2013 Mar 18;8:42. doi: 10.1186/1750-1172-8-42. PMID 23497636